CLINICAL TRIAL: NCT01574196
Title: Assessment of Cardiac Autonomic Function in Adulthood After Chemotherapy or Radiotherapy in Childhood. Ancillary Study of the "Long-term Follow-up of Childhood Cancer Survivors in the Rhône-Alpes and Auvergne Regions of France" Study
Brief Title: Assessment of Cardiac Autonomic Function in Adulthood After Chemotherapy or Radiotherapy in Childhood
Acronym: SALTO-SNA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1108162; 2011-A01357-34 (Other: AFSSAPS)
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Cancer; Sequels; Complications; Autonomic Nervous System
Keywords: Childhood cancer; Cancer; Sequels; Complications; Chemotherapy; Radiotherapy; Surgery; Autonomic nervous system; Parasympathetic Nervous System; Sympathetic Nervous System
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young adult survivors of childhood cancer: Young adult survivors of childhood cancer diagnosed between 1987 and 1992 in the Rhône-Alpes and Auvergne regions of France.
  Interventions: Other: Autonomic nervous system activity records

INTERVENTIONS:
Other: Autonomic nervous system activity records — The description of autonomic equilibrium is based on the use of non-invasive tools such as Holter-ECG monitor (24 hours) which is suitable for longitudinal follow up of cohorts of patients. This tool allows the analysis of instantaneous or delayed variability of the heart rate, in the Hertzian frequency domain after extraction and mathematical transformation of a temporal sequence of R-R spaces from the ECG signal.

SUMMARY:
The SALTO-SNA study is an ancillary study of the SALTO study (Suivi À Long Terme en Oncologie des enfants guéris d'un cancer pédiatrique en régions Rhône-Alpes et Auvergne) coordinated by Dr. Claire Berger, pediatric oncologist at the CHU, Saint Etienne. It aims at re-examining, in their initial treatment center, all patients (a cohort of 495 patients alive in 2011), diagnosed between 1987 and 1992, and cured of childhood cancer (except leukemia) in the Rhône-Alpes and Auvergne regions.

The rationale for this study is based on the observation that although the survival rate of childhood cancers has now reached 75%, complications of chemotherapy and radiotherapy are high and greatly increase the risk of mortality in later years (estimated to be 14% in the literature).

The morbidity risk of chemotherapy and radiotherapy can be quantified by assessing the activity of the intrinsic cardiac autonomic regulation, which represents a powerful predictor of cardiovascular morbidity to the individual.

DETAILED DESCRIPTION:
For this purpose, analysis of the cardiac RR variability is a reliable, non-invasive and reproducible system that could be used in this population as a tool for early detection of cardiovascular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Included in the SALTO study
* Having signed the informed consent form

Exclusion Criteria:

* General anesthesia in the two weeks prior to recording
* Known allergy to electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort study in non-leukemia cancer survivors diagnosed between 1987 and 1992 in the Rhône-Alpes and Auvergne regions of France, who were younger than 15 years at the time of diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Autonomic nervous system activity | 15 years after the end of the cancer treatment
  The autonomic status will be classified in sympatho-vagal equilibrium as "normal", "altered" or "severely abnormal" according to the values obtained for some temporal indices (SDNN, SDaNN, RMSSD etc. ..) and frequencies (Ptot, HF, LF , VLF, ratio LF / HF) compared to validated standards for the age (mean +/- standard deviation).

SECONDARY OUTCOMES:
Doses of radiotherapy | 15 years after the end of the cancer treatment
  Regarding radiotherapy, the doses of different vital organs of the body (151 anatomic sites) will be estimated from the radiotherapy technical records with the help of the Dos-EG software proposed by the INSERM team of F De Vathaire.

CONTACTS AND LOCATIONS:
Overall Officials: Claire BERGER, MD, Principal Investigator — CHU de Saint-Etienne; Hugues PATURAL, MD PhD, Study Director — CHU de Saint-Etienne
Locations (4):
- France (4):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - IHOP, Lyon
  - CHU de Saint-Etienne, Saint-Etienne